CLINICAL TRIAL: NCT03679442
Title: Macrophage Activation, Assessed by Macrophage Markers Soluble CD163 and Soluble CD206, as Indication of Early Liver Cell Damage in Paracetamol Overdose
Brief Title: Macrophage Markers, Soluble CD163 (sCD163) and Soluble CD206 (sCD206) in Paracetamol Overdose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Council for Strategic Research (Other); Novo Nordisk A/S (Industry); Savværksejer Jeppe Juhl og Hustru Ovita Juhls mindelegat (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PCMsCD163NAC
Record Dates: First submitted 2018-09-17; First posted 2018-09-20 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Drug-Induced Acute Liver Injury
Keywords: macrophage activation, N-acetylcysteine, acetaminophen
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy individuals (Experimental): Healthy individuals received intravenous N-acetylcysteine (NAC) treatment to investigate its actions on macrophage activation assessed by the markers soluble CD163 and CD206
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — Non-randomized exposure to N-acetylcysteine (NAC) of healthy individuals corresponding to the clinical treatment guidelines for paracetamol-overdosed patients
  Other Names: NAC; Paracetamol antidote; Acetylcysteine

SUMMARY:
Paracetamol (PCM) is a widely used over-the-counter analgesic, and overdose with PCM is a condition regularly seen in everyday clinical practice. Identification of the patients with early signs of liver injury that may develop into acute liver failure is important. Previous research has shown that macrophages play a role in the development of liver damage in PCM-induced acute liver failure, making macrophage markers interesting possible biomarkers of this condition. In the present study, the investigators aimed to investigate the extent and timing of macrophage activation in PCM-induced liver injury by measuring levels of macrophage markers sCD163 and sCD206 in patients admitted with PCM overdose. The investigators also hoped to find out whether these markers are valuable as prognostic markers of severe outcome in these patients.

Furthermore the investigators examined the possible effect of antidote treatment with N-acetylcysteine on activation and function of macrophages by administering NAC to healthy subjects and measuring levels of sCD163 and sCD206 prior to and after completion of treatment.

DETAILED DESCRIPTION:
The part of the study concerning the patients with PCM overdose was strictly observational with measurement of macrophage markers and no other intervention than the NAC treatment administered in the setting of management of the participants PCM overdose according to best clinical practice.

The interventional part of the study which is submitted for registration here concerns only healthy controls who were exposed to NAC treatment in order to assess the direct effects of NAC on macrophages. The participants received NAC treatment according to the same protocol as the PCM overdosed patients, and macrophage activation markers were measured prior to and after 16 hours of NAC treatment. Thus, the involvement of the participants in the study was limited to the 16 hours of NAC treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75

Exclusion Criteria:

* A history of previous illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2015-06-14 (Actual); Study Completion 2017-02-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sCD163 | 16 hours
  Change in macrophage activation marker soluble CD163 after treatment of healthy individuals with N-acetylcysteine
Change from baseline in sCD206 | 16 hours
  Change in macrophage activation marker soluble CD206 after treatment of healthy individuals with N-acetylcysteine

CONTACTS AND LOCATIONS:
Overall Officials: Henning Grønbæk, Principal Investigator — Department of Hepatology and gastroenterology, Aarhus University Hospital